CLINICAL TRIAL: NCT04203329
Title: A Multi-center, Prospective, Single Arm Registry to Evaluate Procedural Outcomes Using the Cardiva VASCADE MVP VVCS Closure Device After Catheter-based Atrial Fibrillation Interventions for Patients Who Are Discharged the Same Day.
Brief Title: AMBULATE Same Day Discharge Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cardiva Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL 0601
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Vascular Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Paroxysmal A-Fib
  Interventions: Device: Femoral Venous Vascular Closure
- Persistent A-Fib
  Interventions: Device: Femoral Venous Vascular Closure
- A-Fib
  Interventions: Device: Femoral Venous Vascular Closure

INTERVENTIONS:
Device: Femoral Venous Vascular Closure — Femoral venous vascular closure following catheter-based cardiac ablation a-fib cases utilizing 6-12 French inner diameter procedural sheaths at time of closure.

SUMMARY:
A multi-center, prospective, single-arm post market registry, designed to collect both performance and complication outcomes when same day discharge is enabled by the study device, in sealing multiple femoral venous access sites at the completion of ablation procedures for atrial fibrillation with or without another arrhythmia, performed through 6 - 12 Fr inner diameter (maximum 15F OD) introducer sheaths.

ELIGIBILITY:
Group 1 Paroxysmal AF

Inclusion Criteria:

Pre-Operative Inclusion:

All subjects are required to meet the following inclusion criteria in order to be considered eligible for participation in this trial:

1. ≥18 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for an elective, non-emergent catheter-based paroxysmal atrial fibrillation ablation procedure with or without another arrhythmia via the common femoral vein(s) using a 6 to 12 Fr inner diameter (max 15F OD) introducer sheath
4. Is accompanied by a person who will be available to assist the subject for 24 hours post-procedure and/or has access to emergency services;
5. Is willing/able to stay overnight at the hospital per physician discretion.
6. Able and willing to complete two follow-up contacts at 2-4 days and 15 (± 5) days post-procedure.
7. Acceptable candidate for emergent vascular surgery, and/or manual compression of the venous access site;

Intra-Operative Inclusion:

All criteria apply:

1. In the Investigator's opinion, the subject is a candidate for Same Day Discharge per protocol (e.g., no new pericardial effusion, post-procedure diuresis not needed, etc.).
2. Physician or designee will be on site for discharge evaluation.
3. Case completed in time for subject to be reasonably recovered and discharged according to protocol.
4. All femoral venous access sites are planned to be closed with the MVP

Note:

Initial subject eligibility will be determined based on pre-operative screening.

Final subject enrollment will be determined at the end the procedure, prior to closure, based on general intra-op exclusion criteria, as well as additional intraoperative criteria. Enrollment is thus determined intra-operatively, at the end of the case and just prior to closure.

Exclusion Criteria:

Pre-Operative Exclusion:

Subjects will be excluded from participating in this study if they meet any of the following criteria prior to initiation of the index procedure:

1. Advanced refusal of blood transfusion, if it should become necessary;
2. Active systemic infection, or cutaneous infection or inflammation in the vicinity of the groin;
3. Pre-existing immunodeficiency disorder and/or chronic use of high dose systemic steroids;
4. Known history of bleeding diathesis, coagulopathy, hypercoagulability, or current platelet count < 100,000 cells/mm3;
5. Severe co-existing morbidities, with a life expectancy of less than 12 months;
6. Currently involved in any clinical trial that may interfere with the outcomes of this study in the opinion of investigator;
7. Femoral arteriotomy in either limb with any of the following conditions:

   1. access within < 10 days
   2. any residual hematoma, significant bruising, or known associated vascular complications
   3. use of a vascular closure device within the previous 30 days;
8. Femoral venotomy in either limb with any of the following conditions:

   1. access within < 10 days
   2. any residual hematoma, significant bruising, or known associated vascular complications
   3. use of a vascular closure device
9. Any planned procedure involving femoral arterial or venous access in either limb within the next 30 days;
10. Any history of deep vein thrombosis, pulmonary embolism or thrombophlebitis;
11. Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
12. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or who are lactating;
13. Extreme morbid obesity (BMI greater than 45 kg/m2) or underweight (BMI less than 20 kg/m2);
14. Unable to routinely walk at least 20 feet without assistance;
15. Known allergy/adverse reaction to bovine derivatives;
16. Administration of low molecular weight heparin (LMWH) within 8 hours before or after the procedure;
17. Planned procedures or concomitant condition(s) that may extend ambulation attempts beyond routine ambulation and/or hospital discharge time (e.g., staged procedure, serious co-morbidity, uncontrolled obstructive sleep apnea, congestive heart failure), in the opinion of the Investigator.
18. Current diagnosis of persistent or permanent atrial fibrillation.

General Intra-op Exclusion Criteria:

Subjects will be excluded from participating in this study if any of the following exclusion criteria occur during the index procedure:

1. Any attempt at femoral arterial access during the procedure;
2. Any procedural complications that may extend routine recovery, ambulation and discharge times;
3. If the physician deems that a different method should be used to achieve hemostasis of the venous access sites, or that the subject should not attempt ambulation according to the protocol requirements;
4. All venous access sites must are subject to the following exclusion criteria, assessed immediately prior to enrollment:

   1. Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, accidental arterial stick with hematoma, "back wall stick", etc.) in any of the study veins;
   2. A procedural sheath < 6 Fr or > 12 Fr in inner diameter is present at time of closure;
   3. Venous access site location is noted to be "high", above the inguinal ligament (cephalad to lower half of the femoral head or the inferior epigastric vein origin from the external iliac vein);
   4. Intra-procedural bleeding around sheath, or suspected intraluminal thrombus, hematoma, pseudoaneurysm, or AV fistula;
   5. Length of the tissue tract, the distance between the anterior venous wall and skin, is estimated to be less than 2.5 cm.

Discharge Evaluation Criteria

1. Physician or designee must perform discharge evaluation.
2. Subject has successfully ambulated without bleeding from access site.
3. Subject has been able to void.
4. No clinically significant ECG findings.
5. Subject is accompanied by a responsible person who will be near them for the next 24 hours. Subjects must meet all Discharge Criteria in order to be eligible for same day discharge at physician discretion.

Group 2 Persistent A-Fib Pre-Operative Inclusion Criteria All subjects are required to meet the following inclusion criteria in order to be considered eligible for participation in this trial:

1. ≥18 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for an elective, persistent atrial fibrillation ablation procedure;
4. Acceptable candidate planned for same day discharge;
5. Able and willing to complete two follow-up contacts at 2-4 days and 15 (± 5) days post-procedure.

Pre-Operative Exclusion Criteria Subjects will be excluded from participating in this study if they meet any of the following criteria prior to initiation of the index procedure:

1. In the index limb(s): Active systemic infection, or cutaneous infection;
2. Known history of bleeding diathesis, coagulopathy, hypercoagulability, or current platelet count < 100,000 cells/mm3;
3. Currently involved in any clinical trial that may interfere with the outcomes of this study in the opinion of investigator;
4. Femoral catheterization procedure in any study limb in the previous 30 days;
5. Any planned procedure involving femoral arterial or venous access in either limb within the next 30 days;
6. History of deep vein thrombosis, pulmonary embolism or thrombophlebitis in the last 12 months;
7. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or who are lactating;
8. Unable to routinely walk at least 20 feet without assistance;
9. Known allergy/adverse reaction to bovine derivatives;
10. Planned procedures or concomitant condition(s) that may extend ambulation attempts beyond routine ambulation and/or hospital discharge time (e.g., staged procedure, serious co-morbidity, uncontrolled obstructive sleep apnea, congestive heart failure, extreme morbid obesity), in the opinion of the Investigator.

Intra-Operative Inclusion Criteria

All criteria apply:

1. In the Investigator's opinion, the subject is a candidate for Same Day Discharge per protocol (no procedure related events/complications e.g., no new pericardial effusion, post-procedure diuresis not needed, etc.).
2. Case completed in time for subject to be reasonably recovered and discharged according to protocol.
3. All femoral venous access sites are planned to be closed with the MVP

Note:

Initial subject eligibility will be determined based on pre-operative screening.

Final subject enrollment will be determined at the end the procedure, prior to closure, based on general intra-op exclusion criteria, as well as additional intraoperative criteria. Enrollment is thus determined intra-operatively, at the end of the case and just prior to closure.

Intra-Operative Exclusion Criteria Subjects will be excluded from participating in this study if any of the following exclusion criteria occur during the index procedure:

1. Any attempt at femoral arterial access during the procedure;
2. In the index limb(s): infection or inflammation in the vicinity of the groin
3. Administration of low molecular weight heparin (LMWH) within 8 hours before or after the procedure;
4. All venous access sites must are subject to the following exclusion criteria, assessed immediately prior to enrollment:

   1. Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, accidental arterial stick with hematoma, "back wall stick", etc.) in any of the study veins;
   2. A procedural sheath < 6 Fr or > 12 Fr in inner diameter is present at time of closure;
   3. Venous access site location is noted to be "high", above the inguinal ligament (cephalad to lower half of the femoral head or the inferior epigastric vein origin from the external iliac vein);
   4. Intra-procedural bleeding around sheath, or forming hematoma at the time of closure;
   5. Length of the tissue tract, the distance between the anterior venous wall and skin, is estimated to be less than 2.5 cm.

Discharge Evaluation Criteria

1. Physician or designee must perform discharge evaluation on the same day as the procedure.
2. Subject has successfully ambulated without bleeding from access site.
3. Subject has been able to void.
4. No clinically significant ECG findings.
5. Subject is accompanied by a responsible person who will be near them for the next 24 hours. Subjects must meet all Discharge Criteria in order to be eligible for same day discharge at physician discretion.

Group 3 All A-Fib Pre-Operative Inclusion Criteria All subjects are required to meet the following inclusion criteria in order to be considered eligible for participation in this trial:

1. ≥18 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for an elective, atrial fibrillation ablation procedure;
4. Acceptable candidate planned for same day discharge;
5. Able and willing to complete two follow-up contacts at 2-4 days and 15 (± 5) days post-procedure.

Pre-Operative Exclusion Criteria Subjects will be excluded from participating in this study if they meet any of the following criteria prior to initiation of the index procedure:

1. In the index limb(s): Active systemic infection, or cutaneous infection;
2. Known history of bleeding diathesis, coagulopathy, hypercoagulability, or current platelet count < 100,000 cells/mm3;
3. Currently involved in any clinical trial that may interfere with the outcomes of this study in the opinion of investigator;
4. Femoral catheterization procedure in any study limb in the previous 30 days;
5. Any planned procedure involving femoral arterial or venous access in either limb within the next 30 days;
6. History of deep vein thrombosis, pulmonary embolism or thrombophlebitis in the last 12 months;
7. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or who are lactating;
8. Unable to routinely walk at least 20 feet without assistance;
9. Known allergy/adverse reaction to bovine derivatives;
10. Planned procedures or concomitant condition(s) that may extend ambulation attempts beyond routine ambulation and/or hospital discharge time (e.g., staged procedure, serious co-morbidity, uncontrolled obstructive sleep apnea, congestive heart failure, extreme morbid obesity), in the opinion of the Investigator.

Intra-Operative Inclusion Criteria

All criteria apply:

1. In the Investigator's opinion, the subject is a candidate for Same Day Discharge per protocol (no procedure related events/complications e.g., no new pericardial effusion, post-procedure diuresis not needed, etc.).
2. Case completed in time for subject to be reasonably recovered and discharged according to protocol.
3. All femoral venous access sites are planned to be closed with the MVP

Note:

Initial subject eligibility will be determined based on pre-operative screening.

Final subject enrollment will be determined at the end the procedure, prior to closure, based on general intra-op exclusion criteria, as well as additional intraoperative criteria. Enrollment is thus determined intra-operatively, at the end of the case and just prior to closure.

Intra-Operative Exclusion Criteria Subjects will be excluded from participating in this study if any of the following exclusion criteria occur during the index procedure:

1. Any attempt at femoral arterial access during the procedure;
2. In the index limb(s): infection or inflammation in the vicinity of the groin
3. Administration of low molecular weight heparin (LMWH) within 8 hours before or after the procedure;
4. All venous access sites must are subject to the following exclusion criteria, assessed immediately prior to enrollment:

   1. Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, accidental arterial stick with hematoma, "back wall stick", etc.) in any of the study veins;
   2. A procedural sheath < 6 Fr or > 12 Fr in inner diameter is present at time of closure;
   3. Venous access site location is noted to be "high", above the inguinal ligament (cephalad to lower half of the femoral head or the inferior epigastric vein origin from the external iliac vein);
   4. Intra-procedural bleeding around sheath, or forming hematoma at the time of closure;
   5. Length of the tissue tract, the distance between the anterior venous wall and skin, is estimated to be less than 2.5 cm.

Discharge Evaluation Criteria

1. Physician or designee must perform discharge evaluation on the same day as the procedure.
2. Subject has successfully ambulated without bleeding from access site.
3. Subject has been able to void.
4. No clinically significant ECG findings.
5. Subject is accompanied by a responsible person who will be near them for the next 24 hours. Subjects must meet all Discharge Criteria in order to be eligible for same day discharge at physician discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ablation procedures for atrial fibrillation with or without another arrhythmia, performed through 6 - 12 Fr inner diameter (maximum 15F OD) introducer sheaths.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
VASCADE MVP VVCS Procedure Success | 1 day
  Patients do not require next day hospital intervention* due to access site-related complications.
Major Complication Rate | 15 Days +/- 5 Days
  On a per-limb basis, the rate of combined major venous access site closure-related complications attributed directly to the closure method within 15 ± 5 days of discharge (i.e., "device-related" with no other likely attributable cause).

SECONDARY OUTCOMES:
Same Day Procedure Success | 1 day
  Patients do not require next day hospital intervention for any procedure-related reason.
Sustained VASCADE MVP VVCS Procedure Success | 15 Days +/- 5 Days
  Patients do not require hospital intervention within 15 days of discharge due to access site-related complications.
Device Success | intra-procedural
  The ability to deploy the delivery system, deliver the collagen, and achieve hemostasis with the VASCADE MVP VVCS.
Minor Complication Rate | 15 Days +/- 5 Days
  On a per-limb basis, the rate of combined minor venous access site closure-related complications attributed directly to the closure method (i.e., "device-related" with no other likely attributable cause.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of Alabama Birmingham, Birmingham, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Coastal Cardiology, San Luis Obispo, California
  - Aurora Denver Cardiology Associates, The Medical Center of Aurora, Aurora, Colorado
  - MedStar Washington, Washington D.C., District of Columbia
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Lahey Clinic, Burlington, Massachusetts
  - Valley Hospital, Ridgewood, New Jersey
  - Wake Med Hospital, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Cardiac Arrhythmia Institute, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Medical City Fort Worth, Fort Worth, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Chippenham Hospital, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No